CLINICAL TRIAL: NCT04576520
Title: Pragmatic Randomized Controlled Trial of Pharmacopuncture Therapy for Chronic Low Back Pain : A Pilot Study
Brief Title: PCT of Pharmacopuncture Therapy for Chronic Low Back Pain : A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS-CT-2020-09
Record Dates: First submitted 2020-09-29; First posted 2020-10-06 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Chronic Low-back Pain
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pharmacopuncture therapy (Experimental): The physicians will choose the type and volume of pharmacopuncture according to participants' conditions.
  Interventions: Procedure: pharmacopuncture therapy
- physical therapy (Active Comparator): The physicians will choose the type and time of physical therapy according to participants' conditions.
  Interventions: Procedure: physical therapy

INTERVENTIONS:
Procedure: pharmacopuncture therapy — This is a pragmatic RCT, so the physicians will choose the type and volume of pharmacopuncture according to participants' conditions.
  Arms: pharmacopuncture therapy
Procedure: physical therapy — This is a pragmatic RCT, so the physicians will choose the type and time of physical therapy according to participants' conditions.
  Arms: physical therapy

SUMMARY:
This is pilot study for a 2-arm parallel pragmatic randomized controlled trial that will compare pharmacopuncture therapy and physical therapy for chronic low back pain.

DETAILED DESCRIPTION:
This is a pragmatic RCT, so the physicians will choose the type and volume of pharmacopuncture and the type and time of physical therapy according to participants' conditions, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. low back pain for more than 6 months
2. Visual Analogue Scale (VAS) of low back pain is more than 5
3. 19-70 years old
4. participants who agreed and wrote informed consents

Exclusion Criteria:

1. Migration of cancer reaching to spine, fracture of spine
2. Progressive neurologic deficits or severe neurologic deficits
3. Cancer, fibromyalgia, RA, or goat
4. Stroke, MI, kidney disease, dimentia, diabetic neuropathy, or epilepsy
5. Participants taking steroid, immunosuppressant, or psychotropic medication
6. Hemorrhagic disease, severe diabetes or taking anticoagulant drug
7. Participants who took NSAIDs or pharmacopuncture within 1 week
8. Pregnant or lactating women
9. Participants who had undergone cervical surgery within 3 months
10. Participants who had participated in other clinical trial within 1 month, or have plan for participation in other trial during follow up period of this trial
11. Participants who can not write informed consent
12. Participants who is difficult to participate in the trial according to investigator's decision

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-03-26 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) of low back pain | Change from baseline VAS at week 6
  Visual analogue scale of low back pain, minimum 0 to maximum 100, which is a higher score means a worse outcome.

SECONDARY OUTCOMES:
Visual analogue scale (VAS) of leg radiating pain | Week 1, 2, 3, 4, 5, 6, 10, 16
  Visual analogue scale of radiating leg pain, minimum 0 to maximum 100, which is a higher score means a worse outcome.
Numeric rating scale (NRS) of low back pain and leg radiating pain | Week 1, 2, 3, 4, 5, 6, 10, 16
  NRS is a pain scale in which the patient indicates their subjective pain as a whole number from 0 to 10, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain and discomfort imaginable'.
Oswestry Disability Index (ODI) | Week 1, 6, 10, 16
  ODI is a functional disability questionnaire. The possible range of each item score is 0 to 5. Total score range is 0 (better outcome) to 100 (worse outcome).
Korean version of the Roland-Morris Disability Questionnaire (RMDQ) | Week 1, 6, 10, 16
  The Roland Morris Disability Questionnaire consists of 24 statements relating to the person's perceptions of their back pain and associated disability. This includes items on physical ability/activity (15), sleep/rest (3), psychosocial (2), household management (2), eating (1) and pain frequency (1). There is no weighting applied to the statements, therefore the score can range from 0 (no disability) to 24 (maximal disability).
Patient Global Impression of Change (PGIC) | Week 6, 10, 16
  Participants rate the improvement after treatment on a 7-point Likert scale (1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.)
Short Form-12 Health Survey version 2 (SF-12 v2) | Week 1, 6, 10, 16
  The SF-12 consists of 12 questions across 8 domains, and higher scores indicate better health-related quality of life.
EuroQol-5 Dimension (EQ-5D-5L) | Week 1, 6, 10, 16
  The EQ-5D-5L consists of 5 questions (mobility, self-care, usual activities, pain, anxiety/depression) that ask about the current state of health, and answers each question with 5 likert. (1=I have no problems about, 2=I have slight problems about, 3=I have moderate problems about, 4=I have severe problems about, 5=I am unable to about)

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, Ph.D, Study Director — Jaseng Medical Foundation
Locations (4):
- South Korea (4):
  - Jaseng Hospital of Korean Medicine, Seoul, Gangnam-Gu
  - Bucheon Jaseng Hospital of Korean Medicine, Bucheon-si, Gyeonggi Province
  - Haeundae Jaseng Hospital of Korean Medicine, Busan
  - Daejeon Jaseng Hospital of Korean Medicine, Daejeon